CLINICAL TRIAL: NCT04592549
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Pharmacokinetics, and Immunogenicity of ADM03820 in Adults
Brief Title: Study of Monoclonal Antibody Cocktail Being Tested for the Prevention of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: Enabling Biotechnologies (EB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADM03820-001
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — ADM03820

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: 150 mg IM injection of active drug or placebo (Experimental): Subjects in cohort 1 will receive a 150 mg dose IM injection of either active drug or placebo.
  Cohort 1 will dose 8 subjects to active drug and 2 subject to placebo
  Interventions: Drug: ADM03820; Other: Placebo
- Cohort 2: 300 mg IM injection of active drug or placebo (Experimental): Subjects in cohort 2 will receive 300 mg IM injection of either active drug or placebo.
  Cohort 2 will dose 8 subjects to active drug and 2 subject to placebo.
  Interventions: Drug: ADM03820; Other: Placebo
- Cohort 3: 300 mg IM injection of active drug or placebo (Experimental): Subjects in cohort 3 will receive 300 mg IM injection of either active drug or placebo.
  Cohort 3 will dose 8 subjects to active drug and 2 subject to placebo
  Interventions: Drug: ADM03820; Other: Placebo
- Cohort 4: 300 mg IM injection of active drug or placebo (Experimental): Subjects in cohort 4 will receive 300 mg IM injection of either active drug or placebo.
  Cohort 4 will dose 8 subjects to active drug and 2 subject to placebo
  Interventions: Drug: ADM03820; Other: Placebo
- Cohort 5: 600 mg IM injection of active drug or placebo (Experimental): Subjects in cohort 5 will receive 600 mg IM injection of either active drug or placebo.
  Cohort 5 will dose 8 subjects to active drug and 2 subject to placebo
  Interventions: Drug: ADM03820; Other: Placebo

INTERVENTIONS:
Drug: ADM03820 — ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
Other: Placebo — Placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, dose escalation study to evaluate the safety, pharmacokinetics, and immunogenicity of ADM03820 administered as IM injections in healthy adults for the prevention of COVID-19.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and tolerability of escalating IM doses of ADM03820 in healthy adults. Secondary objectives include assessing the pharmacokinetic characteristics and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent understood and signed
2. Healthy male or healthy, non-pregnant, non-lactating female
3. Willingness to comply and be available for all protocol procedures for the duration of the study
4. Between the ages of 18 and 55, inclusive on the day of dosing
5. Body Mass Index (BMI) of ≥18.5 and ≤35 kg/m2
6. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test on Day 1 prior to dosing.

   * Note: A woman is considered of childbearing potential unless post-menopausal (> or = 1 year without menses without other known or suspected cause and appropriately elevated FSH) or surgically sterilized via bilateral oophorectomy or hysterectomy
7. Females of childbearing potential and males agree to use acceptable contraception for the duration of the study

   * Note: These include progestin implants, intrauterine devices (IUDs), surgical (hysterectomy or tubal ligation; vasectomy) or abstinence. Use of methods such as progestin injectables, combined oral hormonal contraceptives, condoms, and diaphragms will not be acceptable when used alone, but they could be considered, if used in combination with another method (for example, a female using combined oral contraceptives if her male partner is sterile, or if she and her non-sterile male partner use a double-barrier method), after consultation with the Ology Bioservices MM. All males will be required to use a barrier method (condoms) for the duration of the study
8. Screening laboratory tests are within normal ranges or outside the normal ranges and considered not clinically significant by the Principal Investigator

   1. If urinalysis by dipstick is abnormal, a complete urinalysis with microscopic evaluation will be performed and the results will supersede the results of the dipstick for blood, glucose, and protein.
   2. Menstruating females failing inclusion criteria due to a positive blood on urine test may be retested following cessation of menses.
   3. Other laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or collection or laboratory error may be repeated once.
9. The urine drug screen is negative
10. Breathalyzer test or blood/saliva alcohol test is negative and subject agrees to abstain from alcohol consumption for a period of 2 days prior to dosing and 2 days prior to any study visit.
11. Agree to minimize risk of SARS-CoV-2 infection.

Exclusion Criteria:

1. History of chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject.
2. Subjects with cardiovascular disease
3. Subjects with diabetes
4. Subjects with pulmonary diseases such as COPD or asthma
5. History of severe allergic reactions of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobins.
6. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds)
7. Clinically significant abnormal electrocardiogram at screening.

   * Note: Clinically significant abnormal ECG results include but not limited to:

   complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained ventricular arrhythmia; sustained atrial arrhythmia; two Premature Ventricular Contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; or any condition deemed clinically significant by a study investigator
   * Incomplete right bundle branch block is not exclusionary if there are no abnormal ECG findings and there is no clinical history or evidence on physical examination to indicate cardiac disease.
8. Positive serology results for HIV, HBsAg, or HCV antibodies
9. Febrile illness with temperature ≥38°C within 7 days of dosing
10. Female subject who is pregnant or breastfeeding
11. Donated blood within 56 days of enrollment
12. Known allergic reactions to any of the study product components present in the formulation or in the processing, as listed in the Investigator Brochure
13. Treatment with another investigational drug within 28 days of dosing
14. Treatment with a monoclonal antibody within 3 months of enrollment
15. Positive serology results for SARS-CoV-2 antibodies (Not applicable for Cohort 5).
16. Positive results from a reverse transcriptase polymerase chain reaction (RT PCR) test for SARS CoV 2
17. Receipt of antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin) or blood transfusion within 6 months or within 5 half-lives of the specific product given
18. Active drug or alcohol use disorder or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
19. Use of H1 antihistamines or beta-blockers within 5 days of dosing
20. Use of any prohibited medication within 28 days prior to screening or planned use during the study period

    * Note: Prohibited medications include immunosuppressives (except Nonsteroidal Anti-Inflammatory Drugs [NSAIDS]); immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); anti-neoplastic agents
21. Any specific condition that in the judgment of the investigator precludes participation because it could affect subject safety
22. Plans to enroll or is already enrolled in another clinical trial that could interfere with safety assessment of the investigational product at any time during the study period

    * Note: Includes trials that have a study intervention such as a drug, biologic, or device
23. Is a study site employee or staff

    * Note: Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators
24. Received an approved COVID-19 vaccine (subjects can receive an approved COVID-19 vaccine after completing their Day 90 visit). For Cohort 5, subjects who received a COVID-19 vaccine within 14 days prior to enrollment are excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - ICON Early Phase Services, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 150 mg IM Injection of Active Drug: Subjects in cohort 1 received a 150 mg dose IM injection of active drug. Cohort 1 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
- Cohort 2: 300 mg IM Injection of Active Drug: Subjects in cohort 2 received a 300 mg IM injection of active drug. Cohort 2 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
- Cohort 3: 300 mg IM Injection of Active Drug: Subjects in cohort 3 received a 300 mg IM injection of either active drug. Cohort 3 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
- Cohort 4: 300 mg IM Injection of Active Drug: Subjects in cohort 4 received a 300 mg IM injection of either active drug. Cohort 4 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
- Cohort 5: 600 mg IM Injection of Active Drug: Subjects in cohort 5 received a 600 mg IM injection of either active drug. Cohort 5 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
- Placebo: Subjects in the placebo group received normal saline. The placebo group will consist of 10 subjects.
  Normal Saline: Normal saline, 0.9% Sodium chloride Injection, US Pharmacopeia [USP]
Period: Overall Study
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug | Cohort 2: 300 mg IM Injection of Active Drug | Cohort 3: 300 mg IM Injection of Active Drug | Cohort 4: 300 mg IM Injection of Active Drug | Cohort 5: 600 mg IM Injection of Active Drug | Placebo
Started | 8 | 8 | 8 | 6 | 8 | 10
Completed | 6 | 7 | 8 | 4 | 6 | 9
Not Completed | 2 | 1 | 0 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 150 mg IM Injection of Active Drug or Placebo: Subjects in cohort 1 received a 150 mg dose IM injection of active drug. Cohort 1 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 2: 300 mg IM Injection of Active Drug or Placebo: Subjects in cohort 2 received a 300 mg IM injection of active drug. Cohort 2 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 3: 300 mg IM Injection of Active Drug or Placebo: Subjects in cohort 3 received a 300 mg IM injection of either active drug. Cohort 3 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 4: 300 mg IM Injection of Active Drug or Placebo: Subjects in cohort 4 received a 300 mg IM injection of either active drug. Cohort 4 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 5: 600 mg IM Injection of Active Drug or Placebo: Subjects in cohort 5 received a 600 mg IM injection of either active drug. Cohort 5 will dose 8 subjects to active drug
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 10 | 48
Age, Customized [Count of Participants; unit: Participants]
  ages 18-55 years | 8 | 8 | 8 | 6 | 8 | 10 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 5 | 3 | 5 | 4 | 25
  Male | 6 | 2 | 3 | 3 | 3 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 4 | 2 | 2 | 15
  Not Hispanic or Latino | 7 | 5 | 5 | 2 | 6 | 8 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 1 | 1 | 1 | 6
  White | 5 | 8 | 7 | 5 | 7 | 8 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 6 | 8 | 10 | 48
Height (cm) [Mean (Standard Deviation); unit: cm] | 173.14 (13.440) | 164.16 (8.750) | 165.76 (7.202) | 166.05 (6.859) | 170.31 (10.502) | 172.46 (8.654) | 168.91 (167.75)
Weight [Mean (Standard Deviation); unit: kg] | 82.64 (15.560) | 77.84 (13.175) | 71.79 (10.707) | 75.72 (17.332) | 88.56 (15.208) | 80.71 (13.984) | 79.75 (14.532)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.50 (3.769) | 28.75 (3.418) | 26.14 (3.802) | 27.25 (4.533) | 30.40 (3.509) | 27.04 (3.971) | 27.84 (3.873)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Serious Adverse Events Following Administration of ADM03820 to the Final Visit
Description: Determine number of SAEs after dosing through the final visit
Time Frame: 540 days for Cohorts 1-4, 365 days for Cohort 5, and up to 540 days for placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 10
Participants | 1 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: The Number of Participants With AEs Following Administration of ADM03820 to the Final Visit
Description: Determine the number of AEs after dosing
Time Frame: 540 days for Cohorts 1-4, 365 days for Cohort 5, and up to 540 days for placebo
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Subjects in the placebo group received normal saline. The placebo group will consist of 10 subjects pooled from cohorts 1-5.
  Normal Saline: Normal saline, 0.9% Sodium chloride Injection, US Pharmacopeia [USP]
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug | Cohort 2: 300 mg IM Injection of Active Drug | Cohort 3: 300 mg IM Injection of Active Drug | Cohort 4: 300 mg IM Injection of Active Drug | Cohort 5: 600 mg IM Injection of Active Drug | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 10
Participants | 7 | 7 | 8 | 2 | 5 | 8

3. Primary Outcome: The Number of Participants With Changes From Baseline in Physical Examination, Vital Signs, and Clinical Safety Laboratory Values Following Administration of ADM03820 to the Final Visit
Description: The number of participants that were includes in this data are those who had clinically significant physical examinations, vital signs, and clinical safety laboratory values following administration of ADM03820 to the final visit.
Time Frame: 540 days
Measure: Number; unit: participants
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 10
participants
  Changes from baseline in physical examination | 0 | 3 | 0 | 0 | 0 | 1
  Changes from baseline in vital signs | 0 | 0 | 0 | 0 | 0 | 0
  Changes from baseline in clinical safety laboratory values | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: The Assessment of Peak Plasma Concentration (Cmax) for Total Antibodies of ADM03820 as Measured by Enzyme-linked Immunosorbent Assay (ELISA) Methods Designed for Total Monoclonal Antibody in the Drug Product (Cohorts 1-2).
Time Frame: pre-dose, 2, 4, 8, and 24 hours post-dose, and on Days 3, 4, 8, 15, 30, 45, 60, 90, 120, 150, 180, and 365
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 8
ng/mL | 17356 [12366.4 to 22346.1] | 51909 [20138.2 to 83679.3]

5. Secondary Outcome: The Assessment of Tmax for Total Antibodies of ADM03820 as Measured by Enzyme-linked Immunosorbent Assay (ELISA) Methods Designed for Total Monoclonal Antibody in the Drug Product (Cohorts 1-2).
Time Frame: pre-dose, 2, 4, 8, and 24 hours post-dose, and on Days 3, 4, 8, 15, 30, 45, 60, 90, 120, 150, 180, and 365
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 8
hours | 1427.81 [0.0 to 3894.799] | 3483.54 [0.0 to 7177.138]

6. Secondary Outcome: The Assessment of the Area Under the Plasma Concentration (AUC(0-t)) for the Total Antibodies of ADM03820 as Measured by Enzyme-linked Immunosorbent Assay (ELISA) Methods Designed for Total Monoclonal Antibody in the Drug Product (Cohorts 1-2).
Time Frame: pre-dose, 2, 4, 8, and 24 hours post-dose, and on Days 3, 4, 8, 15, 30, 45, 60, 90, 120, 150, 180, and 365
Measure: Mean (95% Confidence Interval); unit: hour(ug/mL)
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 8
hour(ug/mL) | 41021 [30100.6 to 51940.8] | 156745 [61880.0 to 251609.7]

7. Secondary Outcome: The Assessment of Peak Plasma Concentration (Cmax) for Each of the Monoclonal Antibodies of ADM03820 as Measured by Enzyme-linked Immunosorbent Assay (ELISA) Methods Designed for Total Monoclonal Antibody in the Drug Product (Cohorts 3-5).
Time Frame: pre-dose, 2, 4, 8, and 24 hours post-dose, and on Days 3, 4, 8, 15, 30, 45, 60, 90, 120, 150, 180, and 365
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 6 | 8
ng/mL
  Monoclonal Antibody: Analyte 2130 | 20180 [12690.9 to 27669.3] | 12693 [8615.5 to 16771.1] | 27120 [20673.7 to 33567.2]
  Monoclonal Antibody: Analyte 2381 | 25478 [13996.0 to 36959.6] | 13812 [10415.4 to 17209.0] | 26049 [21916.8 to 30181.0]

8. Secondary Outcome: The Assessment of Tmax for Each of the Monoclonal Antibodies of ADM03820 as Measured by Enzyme-linked Immunosorbent Assay (ELISA) Methods Designed for Total Monoclonal Antibody in the Drug Product (Cohorts 3-5).
Time Frame: pre-dose, 2, 4, 8, and 24 hours post-dose, and on Days 3, 4, 8, 15, 30, 45, 60, 90, 120, 150, 180, and 365
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 6 | 8
hours
  Monoclonal Antibody: Analyte 2130 | 1336.94 [182.378 to 2491.497] | 371 [84.220 to 659.507] | 654.15 [0.0 to 1455.348]
  Monoclonal Antibody: Analyte 2381 | 1510.85 [438.671 to 2583.029] | 371.86 [84.220 to 659.507] | 741.06 [0.000 to 1535.152]

9. Secondary Outcome: The Assessment of Area Under the Plasma Concentration (AUC(0-t)) for Each of the Monoclonal Antibodies of ADM03820 as Measured by Enzyme-linked Immunosorbent Assay (ELISA) Methods Designed for Total Monoclonal Antibody in the Drug Product (Cohorts 3-5).
Time Frame: pre-dose, 2, 4, 8, and 24 hours post-dose, and on Days 3, 4, 8, 15, 30, 45, 60, 90, 120, 150, 180, and 365
Measure: Mean (95% Confidence Interval); unit: hour(ug/mL)
Arm/Group | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 6 | 8
hour(ug/mL)
  Monoclonal Antibody: Analyte 2130 | 50012 [22236.6 to 77788.1] | 25185 [12078.9 to 38290.8] | 71182 [34399.5 to 107965.4]
  Monoclonal Antibody: Analyte 2381 | 65725 [30277.7 to 101172.3] | 32594 [13117.2 to 52071.2] | 79138 [40378.4 to 117897.2]

10. Secondary Outcome: Presence of Anti-drug Antibody (ADA) Levels
Description: This outcome looks at the total number of participants who had ADA levels at each time point
Time Frame: pre-dose, and Day 15, 30, 45, 60, 90, 120, 150, and 180
Measure: Number; unit: participants
Groups:
- Cohort 1: 150 mg IM Injection of Active Drug or Placebo: Subjects in cohort 1 will receive a 150 mg dose IM injection of either active drug or placebo.
  Cohort 1 will dose 8 subjects to active drug and 2 subject to placebo
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 2: 300 mg IM Injection of Active Drug or Placebo: Subjects in cohort 2 will receive 300 mg IM injection of either active drug or placebo.
  Cohort 2 will dose 8 subjects to active drug and 2 subject to placebo.
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 3: 300 mg IM Injection of Active Drug or Placebo: Subjects in cohort 3 will receive 300 mg IM injection of either active drug or placebo.
  Cohort 3 will dose 8 subjects to active drug and 2 subject to placebo
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 4: 300 mg IM Injection of Active Drug or Placebo: Subjects in cohort 4 will receive 300 mg IM injection of either active drug or placebo.
  Cohort 4 will dose 8 subjects to active drug and 2 subject to placebo
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
- Cohort 5: 600 mg IM Injection of Active Drug or Placebo: Subjects in cohort 5 will receive 600 mg IM injection of either active drug or placebo.
  Cohort 5 will dose 8 subjects to active drug and 2 subject to placebo
  ADM03820: ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
  Placebo: Placebo
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8
participants
  Pre-dose | 2 | 0 | 0 | 0 | 1
  Day 15 | 1 | 0 | 0 | 1 | 0
  Day 30 | 1 | 0 | 0 | 0 | 0
  Day 45 | 1 | 0 | 0 | 0 | 0
  Day 60 | 1 | 0 | 0 | 0 | 0
  Day 90 | 2 | 0 | 1 | 0 | 0
  Day 120 | 1 | 0 | 5 | 0 | 0
  Day 150 | 2 | 4 | 2 | 0 | 0
  Day 180 | 3 | 3 | 1 | 0 | 0

11. Secondary Outcome: The Number of Participants With SARS-CoV-2 RT-PCR Positive Symptomatic Illness Occurring After Dosing
Time Frame: 365 days
Measure: Number; unit: participants
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 10
participants
  Visit 1-7 (1-15 days) | 0 | 0 | 0 | 0 | 0 | 0
  Visit 8-9 (30-45 days) | 0 | 0 | 0 | 0 | 0 | 0
  Visit 10 (60 days) | 0 | 0 | 0 | 0 | 0 | 0
  Visit 11 (90 days) | 0 | 0 | 0 | 0 | 0 | 0
  Visit 12 (120 days) | 0 | 0 | 0 | 0 | 0 | 0
  Visit 13 (150 days) | 0 | 0 | 0 | 0 | 0 | 0
  Visit 14 (180 days) | 2 | 1 | 0 | 0 | 0 | 0
  Visit 15 (365 days) | 3 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: The Number of Participants With SARS-CoV-2 RT-PCR Positive Severe or Critical Symptomatic Illness Occurring After Dosing
Time Frame: 365 days
Measure: Number; unit: participants
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: The Number of Participants With COVID-19 Related Emergency Department Visits Occurring After Dosing
Time Frame: 365 days
Measure: Number; unit: participants
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: The Presence of Neutralizing Antibody Concentrations of ADM03820 as Measured by Microneutralization (MN) Methods
Time Frame: 180 days
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 8
ng/mL
  Pre-dose | 117.0 [NA to NA] — below the level of detection | 117.0 [NA to NA] — below the level of detection | 117.0 [NA to NA] — below the level of detection | 130.6 [98.5 to 173.1] | 1864.4 [937.8 to 3706.7]
  Day 2 | 1840.8 [905.9 to 3740.4] | 1209.1 [635.4 to 2300.8] | 1113.9 [373.6 to 3320.9] | 470.6 [290.9 to 761.3] | 2469.4 [1342.8 to 4541.2]
  Day 15 | 2917.7 [1945.0 to 4376.9] | 3135.1 [2079.3 to 4727.2] | 4340.8 [2880.1 to 6542.1] | 1759.7 [1346.7 to 2299.2] | 3593.4 [2249.8 to 5739.4]
  Day 30 | 3024.5 [1839.6 to 4972.6] | 4835.5 [2367.3 to 9877.1] | 3135.1 [2394.3 to 4105.1] | 1613.5 [1327.1 to 1961.7] | 3020.3 [1695.6 to 5379.8]
  Day 60 | 1149.1 [782.5 to 1687.4] | 3419.0 [2209.2 to 5291.2] | 2543.2 [1925.4 to 3359.3] | 1223.1 [600.0 to 2493.0] | 3135.2 [1716.5 to 5726.5]
  Day 90 | 1748.3 [931.0 to 3283.2] | 2113.3 [918.7 to 4861.4] | 918.3 [500.4 to 1685.5] | 806.9 [487.2 to 1336.4] | 3692.0 [1609.8 to 8467.4]
  Day 120 | 800.2 [415.5 to 1543.0] | 767.9 [436.9 to 1349.5] | 1510.1 [1039.5 to 2193.7] | 595.9 [348.2 to 1019.8] | 3450.7 [1507.1 to 7900.6]
  Day 150 | 230.6 [155.4 to 342.2] | 1424.9 [640.1 to 3171.6] | 1108.9 [690.5 to 1780.8] | 554.4 [209.1 to 1469.7] | 2488.5 [1068.0 to 5798.6]
  Day 180 | 579.0 [339.1 to 988.4] | 690.5 [220.4 to 2163.4] | 784.2 [338.9 to 1814.6] | 421.3 [334.5 to 530.6] | 2173.8 [973.7 to 4852.7]

ADVERSE EVENTS:
Time Frame: 540 days for Cohorts 1-4, including placebo subjects and 365 days for Cohort 5, including placebo subjects
Groups:
- Placebo: Subjects in the placebo group received normal saline. The placebo group consisted of 10 subjects pooled from Cohorts 1-5.
  Normal Saline: Normal saline, 0.9% Sodium chloride Injection, US Pharmacopeia [USP]
Arm/Group | Cohort 1: 150 mg IM Injection of Active Drug or Placebo | Cohort 2: 300 mg IM Injection of Active Drug or Placebo | Cohort 3: 300 mg IM Injection of Active Drug or Placebo | Cohort 4: 300 mg IM Injection of Active Drug or Placebo | Cohort 5: 600 mg IM Injection of Active Drug or Placebo | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 0/8 | 0/6 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8 | 8/8 | 2/6 | 5/8 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 150 mg IM Injection of Active Drug or Placebo (N=8) | Cohort 2: 300 mg IM Injection of Active Drug or Placebo (N=8) | Cohort 3: 300 mg IM Injection of Active Drug or Placebo (N=8) | Cohort 4: 300 mg IM Injection of Active Drug or Placebo (N=6) | Cohort 5: 600 mg IM Injection of Active Drug or Placebo (N=8) | Placebo (N=10)
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chronic Inflammatory Demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arterial Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 150 mg IM Injection of Active Drug or Placebo (N=8) | Cohort 2: 300 mg IM Injection of Active Drug or Placebo (N=8) | Cohort 3: 300 mg IM Injection of Active Drug or Placebo (N=8) | Cohort 4: 300 mg IM Injection of Active Drug or Placebo (N=6) | Cohort 5: 600 mg IM Injection of Active Drug or Placebo (N=8) | Placebo (N=10)
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 1 | 0 | 1 | 3
Activate partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0
Granulocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Mean platelet volume increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Red cell distribution width decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Blood creatinine abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood pressure systolic abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood urea abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Nitrite urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Red blood cell count abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
White blood cell count abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Activate partial thromboplastin time abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin unconjugated decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT04592549/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT04592549/SAP_001.pdf